CLINICAL TRIAL: NCT01897844
Title: A Two-part Phase I Study in Male Healthy Volunteers to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Repeated Incremental Doses of ITF2984. Part A is Double-Blind, Randomized, Subcutaneous Administration. Part B is Open Label, Continuous Infusion.
Brief Title: A Two Part Phase 1, Repeated Doses and Continuous Infusion Study With ITF2984 in Healthy Volunteers
Acronym: 14 days MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSC/13/2984/03; 2013-001076-38 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ITF2984/Placebo 2000 mcg sc bid (Experimental): ITF2984/Placebo 2000mcg s.c. b.i.d. for 14 days
  Interventions: Drug: ITF2984 (100, 2000, 3000 mcg bid); Drug: Placebo
- ITF2984/Placebo 3000 mcg sc bid (Experimental): ITF2984/Placebo 3000mcg s.c. b.i.d. for 14 days
  Interventions: Drug: ITF2984 (100, 2000, 3000 mcg bid); Drug: Placebo
- ITF2984/Placebo 100 mcg sc bid (Experimental): ITF2984/Placebo 100mcg s.c. b.i.d. for 14 days
  Interventions: Drug: ITF2984 (100, 2000, 3000 mcg bid); Drug: Placebo

INTERVENTIONS:
Drug: ITF2984 (100, 2000, 3000 mcg bid)
  Other Names: somatostatin analogues
Drug: Placebo

SUMMARY:
The purpose of this study is to assess the safety,tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of an extended dosing regimen of ITF2984: part A, designed as double-blind, placebo-controlled, randomized, tested an extended dosing regimen, i.e. 14 consecutive dosing days and higher doses, i.e. up to 6000 mcg/day and in part B, open label, continuous subcutaneous infusion for 7 days were tested as ascending doses of ITF2984 up to 9000 mcg/day of ITF2984.

DETAILED DESCRIPTION:
This was a two part Phase I repeated incremental doses study in male healthy volunteers. The study was conducted in two parts. A total of 36 subjects was planned to be enrolled in Part A and 36 subjects in Part B. Part A was performed according to a double blind, randomized, placebo controlled design and included three sequential dose groups of repeat doses. Each group enrolled 12 subjects on ITF2984 or placebo (ratio 9 active: 3 placebo) and received ITF2984 s.c. or placebo twice daily for 14 days. For all three groups the last dose was planned to be the first dose on Day 14.

The study started with the Group 1 2000mcg s.c. b.i.d., Group 2 received 3000mcg b.i.d. after an interim review of the safety and PK data of the 2000mcg dose level. Group 3 received 100mcg s.c. to gather data to complete the PK/PD profile of ITF2984. Subjects were screened up to 28 days before dosing with ITF2984/placebo that took place on Days 1-14.

For all Groups, on day -1 and day 13 subjects received the exogenous tests administration (GHRH, Arginin and TRH) 30 minutes after the first morning administration of ITF2984/placebo.

Part B was open label, and planned for six sequential dose groups of 6 subjects each. In each group subjects received ITF2984 continuous subcutaneous infusion for 7 consecutive days. The dose was escalated, from the starting dose of 900 mcg, by a maximum of three fold or more cautiously, if deemed necessary. The decision to test higher dose levels was based on review of safety and PK data from the previous dose level(s). After a 28 day screening period, subjects were admitted to the clinical unit on the evening of day -2. ITF2984 continuous infusion planned from day 1 to day 8 in the morning. On day -1 (the day prior to the start of infusion) subjects received the exogenous/challenge test administrations (GH-RH+Arginina and TRH). On day 7 the challenge tests were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged 18 to 55 y.o., inclusive, at the time of signing the informed consent
* Body Mass Index (BMI) of 18 to 25 kg/m2, inclusive
* Must be willing and able to communicate and participate in the whole study
* An understanding, ability and willingness to fully comply with study procedures and restrictions.
* Ability to provide written, personally signed and dated informed consent to participate in the study before completing any study-related procedures.
* Subject must be willing to comply with any applicable contraceptive requirements of the protocol
* Satisfactory medical assessment with no clinically significant or relevant abnormalities in the current medical conditions, physical examination, vital signs, ECG and laboratory evaluation as assessed by the Investigator

Exclusion Criteria:

* Current or recurrent disease that could affect the action, absorption or disposition of the investigational medicinal product, or could affect clinical or laboratory assessments.
* Current or relevant previous history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the IMP or study procedures.
* History or presence at the moment of screening visit of gallstones.
* Significant illness, as judged by the Investigator, within 2 weeks of the first dose of IMP.
* Use of prescription or non-prescription drugs (other than 2 g per day paracetamol), including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Known or suspected intolerance or hypersensitivity to the IMP, closely related compounds or any of the stated ingredients.
* History of regular alcohol consumption within 6 months of the study
* A positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* A positive test for HIV antibody.
* Current use of tobacco or other nicotine containing products in any form. Ex users must report that they have stopped using tobacco for at least 90 days prior to receiving the first dose of investigational medicinal product.
* A breath carbon monoxide reading of greater than 10 ppm at screening.
* Any condition that results in a whole blood loss greater than 500 mL within a 90 days period before study participation.
* The subject has participated in a clinical trial and has received an investigational product within the 6 months prior to the first dosing day in the current study(rescreening for subjects that does not have received the study drug during this study is allowed).
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the Investigator.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated
* Subjects fail to satisfy the Investigator of his fitness to participate in this study for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To investigate the safety profile of repeated doses of ITF2984 | 15 days
  Adverse events; 12-lead ECG, including QTc; vital signs (blood pressure, heart rate and body temperature); clinical laboratory evaluations (haematology, clinical chemistry including peripheral glucose, urinalysis), gallbladder volume evaluation.
To investigate the pharmacokinetics (PK) profile of multiple ascending doses of ITF2984 | 15 days and day 8
  Plasma concentrations of ITF2984
To investigate the safety profile of repeated doses of ITF2984 | 8 days
  Adverse events; 12-lead ECG, including QTc; vital signs (blood pressure, heart rate and body temperature); clinical laboratory evaluations (haematology, clinical chemistry including peripheral glucose, urinalysis.

SECONDARY OUTCOMES:
To investigate the effects of ITF2984 on growth hormone (GH) after exogenous growth hormone releasing hormone (GH-RH) and arginine stimulus | 13 Days and 7 Days
  PD biomarkers of GH
To investigate the effects of ITF2984 on thyroid stimulating hormone (TSH) after exogenous thyrotrophin releasing hormone (TRH) stimulus | 13 days and 7 days
  PD biomarkers of TSH
To investigate the effects of ITF2984 on IGF-1 | 13 days and 7 days
  PD biomarkers of IGF-1
To investigate the effects of ITF2984 on glucose | 14 days and 6 days
  PD biomarkers of glucose
To investigate the effects of ITF2984 on prolactin (PRL) after exogenous thyrotrophin releasing hormone (TRH) stimulus | 13 days and 7 days
  PD biomarkers of PRL
To investigate the effects of ITF2984 on insulin | 14 days and 6 days
  PD biomarkers of insulin
To investigate the effects of ITF2984 on glucagon | 14 days and 6 days
  PD biomarkers of glucagon

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ziviani, MD, Principal Investigator — Centro Ricerche Cliniche Verona
Locations (1):
- Centro Ricerche Cliniche, Verona, Verona, Italy